CLINICAL TRIAL: NCT07253675
Title: Phase 2 Double-Blind, Randomized, Controlled Study of MVA-SIBP Vaccine for Mpox in Age De-escalation in the Democratic Republic of the Congo
Brief Title: Evaluate the Safety and Immunogenicity of the MVA-SIBP Vaccine in the Democratic Republic of the Congo
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Institute Of Biological Products (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SIBP-V08-02
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-10

CONDITIONS: Monkeypox (Mpox)
Keywords: Monkeypox; vaccine; safety; immunogenicity
MeSH Terms: conditions — Mpox, Monkeypox | interventions — smallpox and monkeypox vaccine modified vaccinia ankara-bavarian nordic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group 1 (Experimental): MVA-SIBP low dose: low dose monkeypox vaccine produced by Shanghai Institute of Biological Products Co., Ltd. (SIBP)
  Interventions: Biological: MVA-SIBP low dose
- Experimental group 2 (Experimental): MVA-SIBP high dose: high dose monkeypox vaccine produced by Shanghai Institute of Biological Products Co., Ltd. (SIBP)
  Interventions: Biological: MVA-SIBP high dose
- Control group (Active Comparator): MVA-BN: monkeypox vaccine produced by Bavarian Nordic(BN)
  Interventions: Biological: MVA-BN

INTERVENTIONS:
Biological: MVA-SIBP low dose — Participants received one subcutaneous dose of 0.5ml MVA-SIBP low dose on days 0 and 28, respectively, for a total of two doses.
  Arms: Experimental group 1
Biological: MVA-SIBP high dose — Participants received one subcutaneous dose of 0.5ml MVA-SIBP high dose on days 0 and 28, respectively, for a total of two doses.
  Arms: Experimental group 2
Biological: MVA-BN — Participants received one subcutaneous dose of 0.5ml MVA-BN low dose on days 0 and 28, respectively, for a total of two doses.
  Arms: Control group

SUMMARY:
To evaluate the safety and immunogenicity of the MVA-SIBP vaccine using a double-blind, randomized, controlled, age de-escalation design conducted in Kinshasa, Democratic Republic of the Congo (DRC).

DETAILED DESCRIPTION:
Given the urgent need for pediatric data and the high burden of mpox in the DRC, this trial will evaluate the safety and immunogenicity of the MVA-SIBP vaccine using a double-blind, randomized, controlled, age de-escalation design conducted in Kinshasa, DRC. The trial is designed to generate critical data to support regulatory approval and broader access to affordable, stable, and scalable mpox vaccines for Africa.

ELIGIBILITY:
Inclusion Criteria:

* Adults: 18 to 45 years inclusive at the time of informed consent. Adolescents: 12 to 17 years inclusive at the time of consent/assent. Children: 2 to 11 years inclusive at the time of consent/assent.
* Participant is in good general health as determined by medical history, targeted physical examination, and clinical judgment of the investigator.
* Adults: Able to read and understand the written informed consent, and willing to comply with all study procedures and availability for the entire study duration. Adolescents: Parent(s) or legally acceptable representative(s) able and willing to provide written informed consent; participant able and willing to provide appropriate assent per local regulations and IRB requirements. Children: Parent(s) or legally acceptable representative(s), with the relationship to the child similarly verified and documented on the consent form, and able and willing to provide written informed consent.
* Willing and able to comply with all study procedures, visit schedule, and follow-up requirements as judged by the investigator.
* No history of smallpox or mpox vaccination. No history of confirmed or suspected infection with monkeypox, cowpox, or vaccinia virus.
* Negative serum or urine pregnancy test at screening and prior to each vaccination. Willing to use highly effective contraception from 30 days prior to first vaccination through 60 days after the last dose. Breastfeeding.
* Resides in the study catchment area and has no plans to relocate for the duration of the study. Has reliable access to a telephone and/or other means of contact.
* Adults must have been born in 1980 or later. Able to provide direct written informed consent.
* Adolescents: Able to provide written or written assent as appropriate. Children: Parent(s)/guardian(s) able to provide written informed consent; child able to provide assent if developmentally appropriate.

Exclusion Criteria:

* Any prior smallpox or mpox vaccination. History of confirmed or suspected infection with monkeypox, cowpox, or vaccinia virus.
* Close contact, as defined by WHO.
* Known or suspected immunocompromised state as specified in the protocol.
* Acute febrile illness (≥38.0°C) or clinically significant infection within 72 hours prior to vaccination. Any acute illness requiring systemic therapy or hospitalization within 14 days prior to enrollment.
* History of severe allergy or anaphylaxis to any vaccine or vaccine component. History of severe allergic asthma or asthmatic reactions.
* Pregnant or breastfeeding at screening or planning to become pregnant during the study period.
* Participation in another clinical trial with an investigational product or vaccine within 6 months prior to enrollment or planned during the study.
* Receipt of any live vaccine within 28 days or inactivated vaccine within 14 days prior to enrollment or planned within 28 days after any study vaccination.
* Any medical disease or condition that, in the opinion of the investigator, would place the participant at unacceptable risk, interfere with study objectives, or compromise protocol compliance.
* Blood transfusion within three months before inclusion. Significant laboratory test result abnormalities should be added as exclusion criteria. Any condition that, in the opinion of the investigator, would preclude safe participation or successful completion of the study.

Ages: 2 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Unsolicited adverse events | Day 28 after each dose
  An unsolicited AE is any AE reported in addition to those solicited during the clinical study.
Solicited local adverse events | Day 8 after each dose
  That is frequency of occurrence of events pain, erythema, swelling, induration, pruritus at injection site and recorded by memory aid.
Solicited systemic adverse events | Day 8 after each dose
  That is frequency of occurrence of events headache, fatigue, myalgia, fever, chills, nausea and recorded by memory aid.
Serious Adverse Events(SAEs) | Day 365 after the first dose
  To evaluate the incidence of SAE after vaccination.
Adverse Events of Special Interest(AESIs) | Day 365 after the first dose
  To evaluate the incidence of AESI after vaccination.
Medically Attended Adverse Events(MAAEs) | Day 365 after the first dose
  To evaluate the incidence of MAAE after vaccination.
Grade 3+ related adverse events | Day 28 after each dose
  Grade 3+ incidence of adverse events related to vaccination.

SECONDARY OUTCOMES:
Plaque Reduction Neutralization Test(PRNT) Geometric Mean Titers(GMT) of vaccinia | Day 0, 28, 56, 181, 365
  Neutralizing antibody titer by PRNT against vaccinia virus.
PRNTest GMTof mpox | Day 0, 28, 56, 181, 365
  Neutralizing antibody titer by PRNT against mpox virus.
Seroconversion rate of vaccinia | Day 28, 56, 181, 365
  Seroconversion rate is ≥4-fold rise in PRNT titer vs. baseline.
Seroconversion rate of mpox | Day 28, 56, 181, 365
  Seroconversion rate is ≥4-fold rise in PRNT titer vs. baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Hypolite Muhindo Mavoko, Principal Investigator — University of Kinshasa

IPD SHARING:
Plan to Share IPD: No